CLINICAL TRIAL: NCT00098540
Title: Phase II Study of the Raf Kinase Inhibitor BAY43-9006 in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Sorafenib in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01818; N0326; NCCTG-N0326; CDR0000398203; U10CA025224 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with stage IIIB or stage IV non-small cell lung cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with stage IIIB or IV non-small cell lung cancer treated with sorafenib.

II. Determine the clinical toxic effects of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the 24-week progression-free survival rate in patients treated with this drug.

II. Determine the overall survival of patients treated with this drug. III. Determine the time to disease progression in patients treated with this drug.

IV. Correlate predictive disease markers (K-ras and B-raf mutations and ERK/pERK, AKT/pAKT, and VEGFR2/p-VEGFR2 expression) in these patients with the activity of this drug.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), meeting 1 of the following stage criteria:

  * Stage IIIB with pleural effusion
  * Stage IV
* Measurable disease

  * At least 1 lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No known brain metastases, even if treated and stable
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* No bleeding diathesis
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (5 times ULN if hepatic metastasis present)
* Creatinine ≤ 1.5 times ULN
* No uncontrolled hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* HIV negative
* Able to swallow tablets
* No uncontrolled infection
* No other severe underlying disease that would preclude study participation
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated noninvasive carcinomas
* No prior immunotherapy, biologic therapy, or gene therapy
* No concurrent prophylactic colony-stimulating factors
* At least 4 weeks since prior low-dose weekly chemotherapy as a radiosensitizer
* No other prior chemotherapy for NSCLC
* No concurrent chemotherapy
* See Chemotherapy
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to ≥ 30% of bone marrow
* No concurrent radiotherapy

  * Concurrent palliative radiotherapy to nontarget lesions (e.g., painful pre-existing bony metastasis) allowed
* Prior adjuvant therapy allowed provided recurrent disease occurred > 6 months after completion of adjuvant therapy
* No prior systemic therapy for NSCLC, including all novel targeted agents (e.g., gefitinib or erlotinib)
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation (e.g., low-dose warfarin) for venous and arterial devices allowed provided PT, INR, and PTT requirements are met
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response according to RECIST criteria | Up to 5 years
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated using the Duffy-Santner approach.

SECONDARY OUTCOMES:
Progression-free survival | At 24 weeks
  The proportion of patients who are progression-free at 24-weeks will be computed and binomial confidence intervals for the true success proportion will be calculated.
Survival time | From registration to death due to any cause, assessed up to 5 years
  Estimated using the method of Kaplan-Meier.
Time-to-disease progression | From registration to documentation of disease progression, assessed up to 5 years
  Estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States